CLINICAL TRIAL: NCT01980407
Title: A Safety and Efficacy Study of S-1, Oxaliplatin, and Leucovorin (SOL) in Patients With Advanced Gastric Cancer
Brief Title: Feasibility Study of SOL (S-1,Oral Leucovorin,and Oxaliplatin) in Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jilin Provincial Tumor Hospital (Other)
Responsible Party: Principal Investigator, Zhang Yue, Head of Department of Integrated Traditional Chinese and Western Medicine, Jilin Provincial Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JPCH1301; TOTMS1311
Record Dates: First submitted 2013-10-27; First posted 2013-11-11 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2013-11

CONDITIONS: Gastric Cancer
Keywords: S-1; Oxaliplatin; Leucovorin; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Leucovorin; Oxaliplatin; Long-Term Synaptic Depression; Formyltetrahydrofolates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOL, single arm (Experimental): S-1 combined with leucovorin and oxaliplatin
  Interventions: Drug: S-1, leucovorin, oxaliplatin

INTERVENTIONS:
Drug: S-1, leucovorin, oxaliplatin — S-1 (20mg), capsule, 40-60mg, bid, p.o., day1-14； Leucovorin (15 mg), tablet, 30mg,Bid, p.o., day1-14; Oxaliplatin (50 mg), injection 85mg/m2, day1.
  Other Names: S-1 (20mg):Taiho Pharmaceutical Co., Ltd.；; formyltetrahydrofolate (15mg); L-OHP (50mg)

SUMMARY:
In China, S-1 is an novel oral fluoropyrimidine with demonstrated high efficacy on gastrointestinal cancer. The new regimen with oxaliplatin and leucovorin is expected to achieve more encouraging efficacy on gastric cancer. This study is aimed to evaluate the feasibility of the SOL regimen on efficacy and tolerability on Chinese patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Histologically or cytologically documented gastric adenocarcinoma
* Performance status (ECOG scale): 0-2
* Life expectancy ≥ 3 months
* No previous treatment(including: radiotherapy,chemotherapy and immunotherapy)
* Prior systemic therapy (for instance, cytotoxic chemotherapy or active/passive immunotherapy) for adjuvant or neoadjuvant treatment for non-metastatic (M0) disease has been completed within 6 months prior to initiation of study treatment.
* WIth Measurable Target lesion
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* History of hypersensitivity to fluoropyrimidines, S-1, oxaliplatin or the ingredients product
* Inadequate hematopoietic function: WBC≦5,000/mm3; ANC≦2,000/mm3; Platelet≦100,000/mm3
* Inadequate organ function which is defined as below:

Total bilirubin >2 pper limit of normal range (ULN); ALT / AST > 2.5 upper limit of normal range (ULN) (>5.0 x ULN if hepatic metastasis); serum creatinine > 2 upper limit of normal range (ULN);

* Symptomatic peripheral neuropathy ≥ NCI CTC AE grade 1;
* Receiving a concomitant treatment with other fluoropyrimidines or fluorocytosine;
* Pregnancy or lactation women, or women with suspected pregnancy or men unless using a reliable and appropriate contraceptive method;
* Mental status is not fit for chemotherapy therapy presence of serious concomitant illness which might be aggravated by study medication;
* History of ventricular arrhythmia or congestive heart failure;
* Active cardiac disease e.g. decompensate myocardial infarction within the 6-month period preceding entry into the study;
* Significant co-morbid medical conditions, including, but not limited to, Chronic obstructive pulmonary disease, interstitial pneumonia ,pulmonary heart failure, renal failure, hepatic failure, haemorrhagic peptic ulcer, mechanical, paralytic or poor control diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6-8 weeks
  Evaluate the objective response rate followed by RECIST 1.1.

SECONDARY OUTCOMES:
Adverse events | 1 year
  Investigators graded all adverse events and toxic effects according to the National Cancer Institute's Common Toxicity Criteria, The number of Participants with adverse events will be recorded at each treatment visit.
Overall survival | 3 year
Progress free survival | up to 9 weeks
  Tumor assessment will be performed every 3 cycles (9 weeks) from the start of treatment until progression or as for the metastatic site developed during the study (including clinical suspicion). In order to confirm objective tumor response, additional confirmatory scan should be obtained at least 4 weeks following the first radiological evidence of tumor response.
Disease control rate | up to 9 weeks
  To Assess disease control rate (DCR) as defined CR + PR + SD assessed by RECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Provincial Tumor Hospital, Changchun, Jilin, China